CLINICAL TRIAL: NCT06844760
Title: Evaluation of Effectiveness and Safety of Stabilized Injectable Hyaluronic Acid (Perleux Body, Produced by Espad Pharmed Company) in the Rejuvenation, Hydration, and Elasticity Improvement of the Neck Area
Brief Title: Evaluation of Effectiveness and Safety of Stabilized Injectable Hyaluronic Acid (Perleux Body, Produced by Espad Pharmed Company) in the Neck Area
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Espad Pharmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PERB.ESP.VL.IV.03
Record Dates: First submitted 2025-02-08; First posted 2025-02-25 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Skin Aging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Perleux body (Experimental)
  Interventions: Device: Hyaluronic Acid (HA)

INTERVENTIONS:
Device: Hyaluronic Acid (HA) — Subjects will be treated with 2cc of Perleux body at baseline. After 4 weeks, a touch-up injection will be performed to achieve optimal improvement.

SUMMARY:
This study aimed to evaluate the safety and effectiveness of stabilized Hyaluronic Acid Injection under the brand name Perleux body for neck skin rejuvenation, elasticity improvement, and hydration enhancement.

Primary objective: Elasticity (R0, R2, and R5) improvement from baseline in neck area at weeks 8 and 16 Hypothesis: Perleux body (produced by Espad Pharmed Co.) has acceptable efficacy and safety profile for neck skin rejuvenation, elasticity improvement, and hydration enhancement.

Secondary objectives: Effectiveness and safety assessment of Perleux body Study design: This is a phase IV, single-arm, and pre-post study Setting: Subjects will be treated with 2cc of Perleux body at baseline. After 4 weeks, a touch-up injection will be performed to achieve optimal improvement.

ELIGIBILITY:
Inclusion Criteria:

* Age between 35 and 60 years (inclusive)
* The presence of visible signs of skin aging, mainly dry neck skin, rough neck skin, loss of elasticity and clear lines and wrinkles (grades 2, 3, and 4 based on the IBSA Neck Laxity Scale)
* Able to follow study instructions and likely to complete all required visits
* Signing the informed consent form and agreeing to the 6-month follow-up

Exclusion Criteria:

* Previous treatment with fillers containing hyaluronic acid in the neck area during the last year
* History of using RF, rejuvenating lasers or intense pulsed light in the last 6 months
* Having systemic diseases that affect skin health, such as vascular collagen diseases, diabetes, hypothyroidism, liver and kidney failure.
* History of systemic use of drugs affecting the skin such as glucocorticoids, isotretinoin, immunomodulators and hormonal drugs in the last 3 months
* History of taking supplements containing collagen, hyaluronic acid and vitamin C in the last 3 months
* History of using topical corticosteroids and retinoids in the last 4 weeks
* Using topical cosmetic products containing anti-aging ingredients in the last 2 weeks
* Pregnant and lactating women
* History of active smoking during the last 2 years
* Major change in lifestyle including diet and physical activities and sun exposure during the study
* History of previous allergy to hyaluronic acid or lidocaine
* Any inflammation, active infection, unhealed old wound, and skin lesions in the injection area
* Using any anticoagulant product, NSAID, or any other drug that increases the risk of coagulation disorders, in the last 7 days
* History of anaphylactic shock
* Being prone to hypertrophic scar formation
* History of autoimmune disease or immune deficiency or using immunosuppressant drugs

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-04 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2024-10-24 (Actual)

PRIMARY OUTCOMES:
Skin elasticity measured with Cutometer | weeks 8 and 16
  Change of elasticity parameters (R0, R2, and R5) at weeks 8 and 16 from the baseline visit

SECONDARY OUTCOMES:
Stratum corneum moisture | weeks 8 and 16
  Change of stratum corneum moisture measured by MPA 580 probes in the neck area at weeks 8 and 16 from the baseline visit
Transepidermal Water Loss (TEWL) | weeks 8 and 16
  Change of TEWL measured by MPA 580 probes in the neck area at weeks 8 and 16 from the baseline visit
General neck condition | weeks 8 and 16
  Improvement in the clear lines and wrinkles of the neck area according to the Institut Biochimique SA (IBSA) Neck Laxity Scale, with grade 1 being normal tissue tone without noticeable laxity and grade 5 being severe laxity with extreme sagging, using before and after photos, by an independent physician
Skin aging | weeks 8 and 16
  Improvement in the clear lines and wrinkles of the neck area according to global aesthetic improvement scale (GAIS), with grade 1 being exceptional improvement and grade 5 being worsened, using before and after photos by an independent physician
Pain intensity | Day 0 and week 4
  Pain intensity using the VAS (visual analogue scale) [from 0 (complete painlessness) to 10 (maximum pain imaginable)].
Participant satisfaction | weeks 8 and 16
  Participant satisfaction by using the VAS [from 0 (complete dissatisfaction) to 10 (complete satisfaction)].
Participant evaluation | weeks 8 and 16
  Evaluation of participants on the improvement of their skin condition in terms of increased hydration, firmness and radiance, by a questionnaire designed by us. The questionnaire consists of five yes-or-no questions.
Safety assessment | Day 0 and weeks 4, 8, 16
  Assessment of adverse events following treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Private Clinic, Tehran, Tehran Province, Iran